CLINICAL TRIAL: NCT00893399
Title: Phase III Study of Chemotherapy in Combination With ATRA With or Without Gemtuzumab Ozogamicin in Patients With Acute Myeloid Leukemia and NPM1 Gene Mutation
Brief Title: Study of Chemotherapy in Combination With All-trans Retinoic Acid (ATRA) With or Without Gemtuzumab Ozogamicin in Patients With Acute Myeloid Leukemia (AML) and Mutant Nucleophosmin-1 (NPM1) Gene Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 09-09
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: adult patients; NPM1 mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): chemotherapy in combination with ATRA with gemtuzumab ozogamicin
  Interventions: Drug: Gemtuzumab Ozogamicin (Mylotarg); Drug: standard chemotherapy
- 2 (Active Comparator): chemotherapy in combination with ATRA without gemtuzumab ozogamicin
  Interventions: Drug: standard chemotherapy

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin (Mylotarg) — Induction Cycle 1, 2: GO 3mg/m² by intravenous infusion (IVI) on day 1 (total dose 3 mg/m2). Start after etoposide IVI. No dose reduction is foreseen in elderly (> 60 yrs) patients.
  Consolidation 1: GO 3mg/m² by intravenous infusion (IVI) on day 1 (total dose 3 mg/m2). Start after first dose of high-dose cytarabine. No dose reduction is foreseen in elderly (> 60 yrs) patients.
  For all patients experiencing prolonged thrombocytopenia CTC-Grade 3/4 during the first or second induction therapy, which occurs for more than day 35 after start of the cycle, the further cycles of therapy will be administered without Gemtuzumab ozogamicin.
  Consolidation 2, 3: no GO
  Arms: 1
Drug: standard chemotherapy — Idarubicin, Etoposide, Cytarabine, ATRA, Pegfilgrastim

SUMMARY:
Randomized Phase-III, two-arm, open-label, multi-center study in adult patients with AML and NPM1 mutation.

Before Amendment No. 4 (December 2013):

Primary Efficacy Objective:

* Evaluation of efficacy based on event-free survival (EFS) after induction and consolidation chemotherapy plus all-trans retinoic acid (ATRA) with or without gemtuzumab ozogamicin (GO) in adult patients with acute myeloid leukemia (AML) and mutant nucleophosmin-1 (NPM1)

After Amendment No. 4 (December 2013):

Primary Efficacy Objective:

* Evaluation of efficacy based on overall survival (OS) after induction and consolidation chemotherapy plus all-trans retinoic acid (ATRA) with or without gemtuzumab ozogamicin (GO) in adult patients with acute myeloid leukemia (AML) and mutant nucleophosmin-1 (NPM1)

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of acute myeloid leukemia according to the World Health Organization (WHO) classification.
* Presence of NPM1 mutation as assessed in one of the central AMLSG reference laboratories.
* Age ≥ 18 years. There is no upper age limit.
* No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis if needed for up to 5 days during the diagnostic screening phase.
* Non-pregnant and non-nursing. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration.
* Female patients in the reproductive age and male patients must agree to avoid getting pregnant or to father a child while on therapy and within one year after the last dose of chemotherapy.

  * Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control: one highly effective method (e.g., IUD, hormonal, tubal ligation, or partner's vasectomy), and one additional effective method (e.g., latex condom, diaphragm, or cervical cap).
  * "Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months.
  * Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy.
* Signed written informed consent.

Exclusion Criteria:

* AML with other recurrent genetic changes (according to WHO 2008):

  * AML with t(8;21)(q22;q22); RUNX1-RUNX1T1
  * AML with inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11
  * AML with t(15;17)(q22;q12); PML-RARA (or other translocations involving RARA)
  * AML with t(9;11)(p22;q23); MLLT3-MLL (or other translocations involving MLL)
  * AML with t(6;9)(p23;q34); DEK-NUP214
  * AML with inv(3)(q21q26.2) or t(3;3)(q21;q26.2); RPN1-EVI1.
* Performance status WHO > 2.
* Patients with ejection fraction < 50% by MUGA or ECHO scan within 14 days of day 1.
* Organ insufficiency:

  * creatinine > 1.5x upper normal serum level
  * bilirubin, AST or ALP > 2.5x upper normal serum level, not attributable to AML
  * heart failure NYHA III/IV
  * severe obstructive or restrictive ventilation disorder.
* Uncontrolled infection.
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
* Known positive for HIV, active HBV, HCV, or Hepatitis A infection.
* Bleeding disorder independent of leukemia.
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-05-12 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | four years

SECONDARY OUTCOMES:
Rates of complete remission after induction therapy (CR) | not later than 56 days
Cumulative incidences of relapse (CIR) and death in CR (CID) | four years
Event-free survival (EFS) | four years
Days in hospital during each cycle and during the whole intervention | 6 months
Type, frequency, severity, timing and relatedness of AEs and laboratory abnormalities observed during different treatment cycles | 6 months
Incidence of infection after induction and consolidation therapy | 6 months
Duration of neutropenia and thrombocytopenia after induction and consolidation therapy | 6 months
Quality of life assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases, late treatment effects, and demographics according to Messerer et al [49] | two years after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Doehner, MD, Principal Investigator — University of Ulm
Locations (60):
- Austria (7):
  - Medizinische Universitäts Graz, Graz
  - Universitätsklinikum Innsbruck, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H., Linz
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Krankenhaus der Elisabethinen Linz, Linz
  - Salzburger Landeskliniken, Salzburg
  - Hanuschkrankenhaus Wien, Vienna
- Germany (53):
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Ubbo-Emmius-Klinik Aurich, Aurich
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Vivantes Klinikum am Urban, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Charité Berlin - Campus Virchow Klinikum, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Darmstadt, Darmstadt
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen Süd, Ev. Krankenhaus Essen-Werden gGmbH, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - St. Franziskus Hospital, Flensburg
  - Klinikum Frankfurt Höchst GmbH, Frankfurt-Höchst
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Universitätsklinikum Gießen, Giessen
  - Wilhelm-Anton-Hospital gGmbH Goch, Goch
  - Universitätsklinikum Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - Klinikum Hanau, Hanau
  - KRH Klinikum Hannover-Siloah, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken GmbH Heilbronn, Heilbronn
  - Universitätskliniken des Saarlandes, Homburg
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Universitätsklinikum Kiel, Kiel
  - Caritas-Krankenhaus Lebach, Lebach
  - Klinikum Lippe-Lemgo, Lemgo
  - Klinikum Lüdenscheid, Lüdenscheid
  - Universitätsklinikum der Otto-von Guericke Universität Magdeburg, Magdeburg
  - Klinikum der Johannes Gutenberg Universität Mainz, Mainz
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum Schwabing, München
  - Klinikum rechts der Isar München, München
  - Lukaskrankenhaus GmbH Neuss, Neuss
  - Ortenau Klinikum Offenburg Gengenbach, Offenburg
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Klinikum Passau, Passau
  - Caritas-Klinik St. Theresia Saarbrücken, Saarbrücken
  - Stauferklinikum Schwäbisch Gmünd, Schwäbisch Gmünd
  - Klinikum Stuttgart - Katharinenhospital, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Helios Klinikum Wuppertal, Wuppertal

REFERENCES:
- [Derived] Miah K, Goeman JJ, Putter H, Kopp-Schneider A, Benner A. Variable Selection via Fused Sparse-Group Lasso Penalized Multi-state Models Incorporating Molecular Data. Biom J. 2025 Dec;67(6):e70087. doi: 10.1002/bimj.70087. PMID 41146443
- [Derived] Dohner H, Weber D, Krzykalla J, Fiedler W, Kuhn MWM, Schroeder T, Mayer K, Lubbert M, Wattad M, Gotze K, Fransecky L, Koller E, Wulf G, Schleicher J, Ringhoffer M, Greil R, Hertenstein B, Krauter J, Martens UM, Nachbaur D, Samra MA, Machherndl-Spandl S, Basara N, Leis C, Schrade A, Kapp-Schwoerer S, Cocciardi S, Bullinger L, Thol F, Heuser M, Paschka P, Gaidzik VI, Saadati M, Benner A, Schlenk RF, Dohner K, Ganser A; German-Austrian AML Study Group. Intensive chemotherapy with or without gemtuzumab ozogamicin in patients with NPM1-mutated acute myeloid leukaemia (AMLSG 09-09): a randomised, open-label, multicentre, phase 3 trial. Lancet Haematol. 2023 Jul;10(7):e495-e509. doi: 10.1016/S2352-3026(23)00089-3. Epub 2023 May 12. PMID 37187198